CLINICAL TRIAL: NCT04863235
Title: Examining the Impact of a Self-compassion Intervention on Physical Activity Behaviour: An Efficacy Trial
Brief Title: Examining the Impact of a Self-compassion Intervention on Physical Activity Behaviour Among People With Prediabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E2020:006E
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: PreDiabetes
Keywords: self-compassion; physical activity; self-regulation; randomized controlled trial; emotions
MeSH Terms: conditions — Prediabetic State; Motor Activity; Self-Control | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The research assistant who is in charge of conducting the statistical analyses will not be involved in the randomization process or running the intervention or control groups.
  Research assistants who will be conducting in-person eligibility and/or follow-up visits (e.g. handing out accelerometers) will be blinded to participant group assignment.
  Participants will also be blinded to which group they are randomized into. The investigators will present the study as examining different education interventions to increase physical activity and will not let the participants know whether they are in the intervention or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Session 1: Participants will meet individually with a research assistant to discuss their type 2 risk, discuss benefits of engaging in 150 minutes of moderate-to-vigorous physical activity per week, and set a physical activity goal. Ideal Care will involve: Session 2: Introductions and Goal setting/planning. Session 3: Monitoring Physical Activity Session 4: Action and Coping Planning. Session 5: Self-Efficacy (master and vicarious experiences). Session 6: Self-Efficacy (modeling experiences, verbal persuasion). Session 7: Physical Activity Enjoyment and Barriers. Session 8: Making long-term Change. The last 30 minutes of sessions 2-6, control participants will receive 30-minutes of non-self-compassion or physical activity related health education (i.e., sleep, screen time, blood pressure, cholesterol, benefits of water, benefits of vitamin D, the Infodemic).
  Interventions: Behavioral: Control Group
- Intervention Group (Experimental): Session 1: Participants will meet individually with a research assistant to discuss their type 2 risk, discuss benefits of engaging in 150 minutes of moderate-to-vigorous physical activity per week and set a physical activity goal. First 30 minutes of each subsequent session will be ideal care (as described above in the control group). Last 30 minutes of sessions 2-6, self-compassion condition participants will learn to apply self-compassion to their prediabetes experience and physical activity. Session 2: Introduction to self-compassion. Session 3: Yin and Yang of self-compassion. Session 4: Mindfulness. Session 5: Mindfulness and Resistance. Session 6: Meeting Difficult Emotions. Session 7: Embracing the Good. Session 8: Applying Self-compassion to Physical Activity and Moving Forward.
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Control Group — Eight week behavioural change program aimed to increase physical activity plus information on general health topics among individuals with prediabetes.
  Arms: Control Group
Behavioral: Intervention Group — Eight week behavioural change program plus a self-compassion intervention aimed to increase physical activity among individuals with prediabetes.
  Arms: Intervention Group

SUMMARY:
The investigators plan to examine whether teaching people at risk for type two diabetes to use self-compassion (orientation to care for oneself during difficult situations) helps them self-manage and increase their physical activity. People at risk for type 2 diabetes will learn about their type 2 diabetes risk and strategies to increase their physical activity, which represents the recommended information that people at risk for type two diabetes should receive. In addition to this, some participants, but not all, will be taught to be self-compassionate in relation to their type two diabetes risk and their efforts to increase their physical activity. The investigators expect that people who receive the additional training about how to be self-compassionate will engage in more physical activity than people who do not and they will do so because of self-compassion's positive effect on aspects of self-management - adaptive reactions and a tendency to use strong self-management skills. This study is important for health promotion because it allows the investigators to determine whether they can improve how they currently help people prevent type 2 diabetes through engaging in physical activity.

DETAILED DESCRIPTION:
The primary research objective of this efficacy trial is to determine if a self-compassion intervention can lead to a clinically significant increase in engagement in physical activity as compared to usual care (best behaviour change practice) in individuals with prediabetes.

Primary research question: Will a self-compassion intervention that augments usual care lead to greater increases in physical activity over 12 weeks post-intervention follow-up than usual care alone among people with prediabetes? Primary hypothesis: Self-compassion will lead to greater increases in physical activity than usual care at intervention-end and at 6- and 12-weeks.

Secondary research question: Will the effects of a self-compassion intervention on physical activity at 6- and 12-weeks post intervention be mediated by (i) negative affect (ii) physical activity self-regulatory skills and (iii) personal growth at baseline and intervention-end? Secondary hypothesis: The effects of self-compassion on physical activity behaviour at 6- and 12-weeks will be mediated by i) affect and ii) self-regulatory skill use assessed at baseline and intervention-end.

Tertiary research question: Will a self-compassion intervention that augments usual care lead to greater increases in other health-promoting behaviours (e.g., nutrition, stress management, seeking medical attention)? Tertiary hypothesis: Self-compassion will lead to greater increases in health-promoting behaviours than usual care at intervention end, 6-weeks and 12-weeks post intervention.

This efficacy trial is a single centre, randomized, active controlled, eight week intervention with baseline and follow-up assessment at intervention-end, 6- and 12-weeks post-intervention. It follows a quantitative-dominant, mixed-methods design. The investigators will compare the change in physical activity of community-dwelling people with prediabetes randomized to usual care in the form of behaviour change + attention (control condition) to that of participants who receive usual care + self-compassion training (intervention condition). The investigators will also examine potential mediators of the intervention (i.e., negative affect, physical activity self-regulatory skill use).

They will supplement this trial with interviews after follow-up testing with a subsample of self-compassion intervention participants. These interviews will provide feasibility information from participants (e.g., receptivity) as well as provide a qualitative assessment of the investigators' outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Medium to high type 2 diabetes risk (assessed with the CANRISK tool)
* Age 40 - 74
* No current medical treatment for type 2 diabetes
* Safe to engage in physical activity
* No non-study self-reported current type 2 diabetes/behaviour change education that may interfere with the intervention
* Available for all sessions and testing
* Insufficient physical activity relative to guidelines of 150 minutes of moderate to vigorous physical activity per week.
* Below the mean on the self-compassion scale

Exclusion Criteria:

* Be under 40 years old, or over the age of 74
* Have a medical condition which would not allow them to participate safely in physical activity
* Already are part of a different behavioural change/ type 2 diabetes education group
* Already engage in over 150 minutes of moderate to vigorous physical activity per week
* Already have high levels of self-compassion (over the mean)
* Could not commit to the intervention/control sessions

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Differences between groups in moderate to vigorous physical activity at 8 weeks | Post-intervention (8 week time point).
  Physical activity as measured by GT3X+ accelerometers (1952 - >9498 counts per min)
Differences between groups in moderate to vigorous physical activity at 14 weeks | 6 week Follow-up (14 week time point)
  Physical activity as measured by GT3X+ accelerometers (1952 - >9498 counts per min)
Differences between groups in moderate to vigorous physical activity at 20 weeks | 12 week Follow-up (20 week time point)
  Physical activity as measured by GT3X+ accelerometers (1952 - >9498 counts per min)
Changes in self-compassion from pre-intervention to post-intervention (8 weeks) | Baseline to Post-Intervention (0 - 8 weeks)
  The Self-Compassion Scale (Neff, 2003a); 26-item scale; assess individuals' current level of self-compassion. The scale has 6 subscales (self-kindness, self-judgment, mindfulness, over-identification, isolation, common humanity. Participants respond to a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always). Subscale means are first calculated and then an overall mean is calculated to give you a total self-compassion score
Changes in self-compassion from pre-intervention to 6 week follow-up (14 weeks) | Baseline to 6 week follow-up (0 - 14 weeks)
  The Self-Compassion Scale (Neff, 2003a); 26-item scale; assess individuals' current level of self-compassion. The scale has 6 subscales (self-kindness, self-judgment, mindfulness, over-identification, isolation, common humanity. Participants respond to a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always). Subscale means are first calculated and then an overall mean is calculated to give you a total self-compassion score
Changes in self-compassion from pre-intervention to 12 week follow-up (20 weeks) | Baseline to 12 week follow-up (0 - 20 weeks)
  The Self-Compassion Scale (Neff, 2003a); 26-item scale; assess individuals' current level of self-compassion. The scale has 6 subscales (self-kindness, self-judgment, mindfulness, over-identification, isolation, common humanity. Participants respond to a 5-point Likert scale ranging from 1 (almost never) to 5 (almost always). Subscale means are first calculated and then an overall mean is calculated to give you a total self-compassion score

SECONDARY OUTCOMES:
Differences between groups in self-reported physical activity at 8 weeks | Post-Intervention (8 week time point)
  Short International Physical Activity Questionnaire (Forde, 2018). 4-item scale; assesses walking, moderate intensity and vigorous intensity activities over the last 7 days.
Differences between groups in self-reported physical activity at 14 weeks | 6 week Follow-up (14 week time point)
  Short International Physical Activity Questionnaire (Forde, 2018). 4-item scale; assesses walking, moderate intensity and vigorous intensity activities over the last 7 days.
Differences between groups in self-reported physical activity at 20 weeks | 12 week Follow-up (20 week time point)
  Short International Physical Activity Questionnaire (Forde, 2018). 4-item scale; assesses walking, moderate intensity and vigorous intensity activities over the last 7 days.
Negative Affect Related to Diabetes at 8 weeks as a potential mediator | Post Intervention (8 week time point)
  Negative Affect Scale (Leary, Tate, Adams, Allen, & Hancock, 2007); 7-point Likert scale ranging from 1 (not at all) to 7 (Extremely); Scale Range: 20 (low Negative Affect) - 140 (high Negative Affect)
Negative Affect Related to Low Physical Activity Engagement at 8 weeks as a potential mediator | Post Intervention (8 week time point)
  Negative Affect Scale (Leary, Tate, Adams, Allen, & Hancock, 2007); 7-point Likert scale ranging from 1 (not at all) to 7 (Extremely); Scale Range: 20 (low Negative Affect) - 140 (high Negative Affect)
Self-regulatory skill use as a potential mediator | Post Intervention (8 week time point)
  Physical activity Self-Regulation scale-12 (Umstattd, Motl, Wilcox, Saunders, & Watford, 2009); 5-point Likert scale ranging from 1 (never) to 5 (very often); Scale Range: 12 (low physical activity self-regulation) - 60 (high physical activity self-regulation)
Differences between groups in health-promoting behaviours at 8 weeks | Post Intervention (8 week time point)
  Health-Promoting Lifestyle Profile II (Walker, Sechrist, & Pender, 1995); 4-point Likert scale ranging from 1 (never) to 4 (routinely); Scale range: 52 (low engagement in health behaviours) to 208 (high engagement in health behaviours)
Differences between groups in health-promoting behaviours at 14 weeks | 6 week Follow-up (14 week time point)
  Health-Promoting Lifestyle Profile II (Walker, Sechrist, & Pender, 1995); 4-point Likert scale ranging from 1 (never) to 4 (routinely); Scale range: 52 (low engagement in health behaviours) to 208 (high engagement in health behaviours)
Differences between groups in health-promoting behaviours at 20 weeks | 12 week Follow-up (20 week time point)
  Health-Promoting Lifestyle Profile II (Walker, Sechrist, & Pender, 1995); 4-point Likert scale ranging from 1 (never) to 4 (routinely); Scale range: 52 (low engagement in health behaviours) to 208 (high engagement in health behaviours)
Differences between groups in seeking medical attention at 8 weeks | Post Intervention (8 weeks)
  Seeking Medical Attention Scale (Terry, Leary, Mehta, & Henderson, 2013); Participants indicate using a yes or no response whether they have sought out medical attention and/or resources (i.e., made a doctor appointment, inquired about community programs, reach out to friend/family member, sought out information, quit smoking, reduced weight)
Differences between groups in seeking medical attention at 14 weeks | 6 weeks Follow-up (14 weeks)
  Seeking Medical Attention Scale (Terry, Leary, Mehta, & Henderson, 2013); Participants indicate using a yes or no response whether they have sought out medical attention and/or resources (i.e., made a doctor appointment, inquired about community programs, reach out to friend/family member, sought out information, quit smoking, reduced weight)
Differences between groups in seeking medical attention at 20 weeks | 12 week Follow-up (20 weeks)
  Seeking Medical Attention Scale (Terry, Leary, Mehta, & Henderson, 2013); Participants indicate using a yes or no response whether they have sought out medical attention and/or resources (i.e., made a doctor appointment, inquired about community programs, reach out to friend/family member, sought out information, quit smoking, reduced weight)
Differences between groups in nutrition at 8 weeks | Post Intervention (8 weeks)
  Dietary Screener Questionnaire; scoring algorithms convert responses to estimates of dietary intake for diary (cup equivalents), fruits and vegetables (cup equivalents), added sugars (tsp), whole grains (ounce equivalents), calcium (mg), fiber (g). Responses to processed meat and red meat questions are used qualitatively as no scoring algorithms are developed for these categories.
Differences between groups in nutrition at 14 weeks | 6 week Follow-up (14 weeks)
  Dietary Screener Questionnaire; scoring algorithms convert responses to estimates of dietary intake for diary (cup equivalents), fruits and vegetables (cup equivalents), added sugars (tsp), whole grains (ounce equivalents), calcium (mg), fiber (g). Responses to processed meat and red meat questions are used qualitatively as no scoring algorithms are developed for these categories.
Differences between groups in nutrition at 20 weeks | 12 week Follow-up (20 weeks)
  Dietary Screener Questionnaire; scoring algorithms convert responses to estimates of dietary intake for diary (cup equivalents), fruits and vegetables (cup equivalents), added sugars (tsp), whole grains (ounce equivalents), calcium (mg), fiber (g). Responses to processed meat and red meat questions are used qualitatively as no scoring algorithms are developed for these categories.
Personal Growth Initiative as a potential mediator | Post Intervention (8 weeks)
  Personal Growth Initiative Scale-II (Robitschek, 2008); 6-point Likert scale ranging from 0 (disagree strongly) to 5 (agree strongly); Scale Range: 0 (low personal growth initiative) - 20 (high personal growth initiative)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada